CLINICAL TRIAL: NCT05044637
Title: Phase IIB Study to Evaluate Primaquine Safety and Tolerability for Radical Cure of Uncomplicated Plasmodium Vivax Malaria in Children < 15 Years-old (CHILDPRIM)
Brief Title: Study to Evaluate Primaquine for Radical Cure of Uncomplicated Plasmodium Vivax Malaria in Children
Acronym: CHILDPRIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 50193921.6.1001.0005
Record Dates: First submitted 2021-08-20; First posted 2021-09-16 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Malaria, Vivax
MeSH Terms: conditions — Malaria, Vivax | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Primaquine (3.5mg x 7d) (Experimental): Primaquine 7 days Standard blood schizontocidal therapy plus 7 days of unsupervised primaquine (3.5 mg/kg total dose) administered once per day (0.5 mg/kg OD).
  Interventions: Drug: Primaquine
- Primaquine (7.0mg x 7d) (Active Comparator): Primaquine 7 days Standard blood schizontocidal therapy plus 7 days of unsupervised primaquine (7.0 mg/kg total dose) administered once per day (1.0 mg/kg OD).
  Interventions: Drug: Primaquine
- Primaquine (7.0mg x 14d) (Active Comparator): Primaquine 14 days Standard blood schizontocidal therapy plus 14 days of unsupervised primaquine (7.0 mg/kg total dose) administered once per day (0.5 mg/kg).
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — 7 days of unsupervised primaquine (3.5 mg/kg total dose) administered once per day (0.5 mg/kg OD).
  Other Names: Low-standard dose
  Arms: Primaquine (3.5mg x 7d)
Drug: Primaquine — 7 days of unsupervised primaquine (7.0 mg/kg total dose) administered once per day (1.0 mg/kg OD).
  Other Names: High-dose short course
  Arms: Primaquine (7.0mg x 7d)
Drug: Primaquine — 14 days of unsupervised primaquine (7mg/kg total dose) administered once per day (0.5 mg/kg).
  Other Names: High-dose long course
  Arms: Primaquine (7.0mg x 14d)

SUMMARY:
The main determinant of primaquine efficacy is the total dose of primaquine administered, rather than the dosing schedule. Infants and children younger than 4 years of age are at a higher risk of frequent relapses than older age groups, which may lead to severe anaemia. In view of this issue, after Glucose-6-phosphate dehydrogenase (G6PD) testing, WHO recommends the use of a low dose (0·25 mg/kg of bodyweight) of primaquine for 14 days in infants aged 6 months and older, as a follow-up treatment for malaria caused by P. vivax and P. ovale. Nevertheless, previous trials have demonstrated that the standard low dose regimen of primaquine (3.5 mg/kg total) fails to prevent relapses in many different endemic locations. For this reason, the 2010 WHO antimalarial guidelines now recommend a high dose regimen of 7 mg/kg (equivalent to an adult dose of 30mg per day), although many countries still recommend lower doses for fear of causing more serious harm to unscreened G6PD deficiency patients.

The pharmacokinetics of several antimalarial drugs are different in children younger than 10 years of age or who are underweight for their age compared with children of 10 years and older and adults.The doses of several antimalarials in children are suboptimal. This oversight is a consequence of designing dosing regimens in a different population (i.e., adults) for the one most affected by the disease and this has led to revisions of some dosing recommendations. The different pharmacokinetic performance of drugs in children might also relate to maturation (e.g., of metabolic processes, particularly in the first 2 years of life). Pharmacogenomic factors affecting drug metabolism are increasingly being studied. Polymorphisms in cytochrome P4502D6 are associated with different primaquine metabolizer phenotypes with resulting differing efficacies for radical cure. Shorter courses of higher daily doses of primaquine have the potential to improve adherence and, thus, effectiveness without compromising efficacy. If the efficacy, tolerability and safety of short-course, high-dose primaquine regimens can be assured across the range of endemic settings, along with reliable point-of-care G6PD deficiency diagnostics, then this would be a major advance in malaria treatment by improving adherence and thus the effectiveness of anti-relapse therapy.

ELIGIBILITY:
Inclusion Criteria:

* Infection with P.vivax parasitaemia;
* ≥ 6 months and ˂ 15 years of age;
* Body weight ≥ 5 Kg;
* Hb > 7 g/dL
* presence of axillary temperature >37.5 Celsius or history of fever during the past 48 hours;
* ability to swallow oral medication;
* Absence of severe malnutrition (defined as a child whose growth standard is below -3-Z-score, has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm)
* Absence of febrile conditions due to disease other than malaria (e.g., measles, acute lower respiratory tract infection, severe diarrhea with dehydration) or the known underlying chronic or severe diseases (e.g., cardiac, renal, hepatic diseases, HIV/AIDS);
* History of hypersensitivity reactions to or contraindicated for any of the medicine(s) being teste d or used as alternative treatment(s);
* A negative pregnancy test or non-lactating
* Ability and willingness to comply with the study protocol for the duration of the study, including 6 months of follow up;
* Informed consent from the patient/parent/guardian (with additional informed assent for any participant between 7 and 14 years of age);
* Pregnancy test consent from girls of childbearing age (defined as having had menarche) and their parents or guardians;

Exclusion Criteria:

* G6PD- Deficiency (< 4.0 U/g Hb)
* The subject has severe P. vivax malaria as defined by the World Health Organization (WHO) criteria
* intolerance of or allergy to one of the medications in the study
* Pregnant or breastfeeding women
* Inability to tolerate oral medication
* Blood tranfusion in the last 3 months (as this may mask the G6PD deficiency)
* Serious or chronic medical condition (cardiac, renal, hepatic diseases, sickle cell disease, HIV/AIDS)
* History of malaria in the last 30 days
* Belonging to the indigenous community

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse Event | 6 months after randomization
  To diagnose, resolve and catalog adverse events of any intensity, whether clinical or laboratory
Efficacy - Radical cure | 6 months after randomization
  The incidence rate (i.e., per person-year) of symptomatic recurrent P. vivax parasitaemia (detected by microscopy) over 6 months of follow-up in the 3.5 mg/Kg total dose versus 7.0 mg/Kg total dose primaquine groups

SECONDARY OUTCOMES:
Incidence rate (per person-year) of recurrent P. vivax | 6 months after randomization
  The overall incidence rate (per person-year) of any recurrent P. vivax parasitaemia detected by microscopy over 6 months of follow-up in the 3.5 mg/Kg total dose group versus the 7.0 mg/Kg total dose groups
Incidence risk of any recurrent symptomatic P. vivax malaria | 6 months after randomization
  The incidence rate (per person-year) of any recurrent symptomatic P. vivax parasitaemia over 6 months of follow-up in either the 7-day or the 14-day primaquine arms of 7.0 mg/kg total dose compared with 7-day primaquine arm of 3.5 mg/Kg total dose.
The hematological recovery in patients with vivax malaria | 6 months after randomization
  Hematological recovery will be assessed as the incidence risk of severe anaemia (Hb<7g/dl) and/or blood transfusion within the 6 month follow up period, and the mean fall in baseline Hb on day 7 and day 14. These outcomes will be compared between the treatment arms
Proportion of patients with any adverse drug reactions | 6 months after randomization
  The proportion of patients with one or more adverse drug reactions within 42 days of their primary treatment and also at 6 months
Primaquine tolerability 1 hour | 7 to 14 days after randomization
  Tolerability of primaquine will be assessed by comparing the proportion of patients with nausea, vomiting, abdominal pain and vomiting of a dose within 1 hour of administration between the treatment arms
Primaquine tolerability | 7 to 14 days after randomization
  Drug tolerability between the treatment arms will also be assessed by comparing the proportion of patients completing a full course of primaquine therapy
Pharmacogenetics CYP2D6 | 1 day after randomization
  Characterize hepatic cytochrome CYP2D6 enzyme phenotypes using Activity Score A (AS-A)
Genotype CYP2D6 | 1 day after randomization
  Genotype CYP2D6 alleles in this study population
Metabolomics | 28 days after randomization
  Describe the metabolic signatures present in patients with adverse events (AEs) and severe AEs (SAEs)

OTHER OUTCOMES:
Exploratory - Pharmacokinetics of primaquine Area Under the Curve (AUC) | 24 hours
  Area under the plasma concentration time AUC 0-∞curve for primaquine and metabolites (mPQ)
Exploratory - Pharmacokinetics of primaquine Conc | 24 hours
  Primaquine and metabolites maximum concentrations
Exploratory - Pharmacokinetics of primaquine Elimination rate | 24 hours
  Primaquine and metabolites (mPQ) elimination rate constants (mPQ-λz)
Exploratory - Pharmacokinetics of primaquine Elimination half-life | 24 hours
  Primaquine and metabolites (mPQ) elimination half- life (mPQ-t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Maria das Graças C Alecrim, PhD, MD, Principal Investigator — Fundação de Medicina Tropical - HVD
Locations (2):
- Brazil (2):
  - Universidade Federal do Acre, Cruzeiro do Sul, Acre
  - Fundação de Medicina Tropical Doutor Heitor Vieira Dourado, Manaus, Amazonas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pacheco ALO, Omena AG, Baia-da-Silva DC, Jardim TAP, Silva DCB, Lopes APB, Barbosa LRA, Souza IG, Araujo RF, Nogueira LOS, Vale SCN, Melo GC, Cordeiro JSM, Bassat Q, Sampaio VS, Lima VDS, Martinez-Espinosa FE, Mourao MPG, Monteiro WM, Alecrim MGC, Brito-Sousa JD, Lacerda MVG. Safety, tolerability, and efficacy of high versus low-dose, short versus long-course daily primaquine for the radical cure of uncomplicated Plasmodium vivax malaria in children under 15 years of age: an open-label, non-inferiority, randomized controlled trial (CHILDPRIM). Malar J. 2025 Dec 22. doi: 10.1186/s12936-025-05686-y. Online ahead of print. PMID 41430686